CLINICAL TRIAL: NCT04188353
Title: Effect of Intravenous Administration of 20% Mannitol on the Optic Nerve Sheath Diameter(ONSD) in Patients With Raised Intracranial Pressure
Brief Title: Effect of Intravenous Administration of Mannitol on ONSD in Patients With Raised ICP
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Shiva Prasad Paudyal, Resident, PGY-III, Anesthesiology, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 360(6-11)E^2/075/76
Record Dates: First submitted 2019-11-09; First posted 2019-12-05 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Raised Intracranial Pressure
Keywords: ONSD; Mannitol; ICP
MeSH Terms: conditions — Intracranial Hypertension | interventions — Mannitol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Optic nerve sheath diameter measurement — ONSD measurements done at screening (T1), 30 minutes after mannitol infusion (T2), 60 minutes (T3) and 120 minutes (T4)
  Other Names: ONSD
Drug: Mannitol — Mannitol at dose of 0.25 to 1 gm/kg over 20 minutes via a dedicated IV line
  Other Names: Osmotherapy

SUMMARY:
Osmotherapy with mannitol has been a common practice in patients with raised ICP. Monitoring its effect on ICP can be performed invasively and non-invasively. Due to a validated correlation between invasive ICP monitoring and ONSD measurement, it can be a tool to monitor acute and long term effects of osmotherapy non-invasively on ICP. This study examines the acute changes in sonographically measured ONSD brought about by the administration of mannitol. This can correlate with the changes in ICP in such patients and can be utilized as a tool for decision making/ point-of-care utility.

DETAILED DESCRIPTION:
This is a prospective cohort based observational study including 40 patients admitted in the adult ICU at our center diagnosed as either a case of TBI/ acute stroke/ intracranial hemorrhages with a mean screening ONSD of more than 5mm under mannitol osmotherapy. ONSD were measured by a high frequency linear array probe (>10 Hz) at the time of screening. Mannitol was then administered at doses prescribed by the treating physician over 20-30 minutes via a dedicated intravenous line. ONSDs were measured again at 30, 60 and 120 minutes after completion of administration of mannitol. Demographic data, baseline ventilator parameters of patients on mechanical ventilation, GCS and mean arterial pressure at each time points were recorded. Comparison of variables at these time points were made.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* diagnosed as a case of TBI/ acute stroke/ intracranial hemorrhages
* screening mean ONSD > 5 mm
* under osmotherapy with mannitol in standard doses (0.25 - 1 gm/kg)

Exclusion Criteria:

* baseline ocular pathology like tumors, Graves' disease and sarcoidosis
* previous ocular surgery
* Decompressive cranial surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Admitted in the ICU of Tribhuvan university teaching hospital within the time period of the study
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-02-24 (Actual); Primary Completion 2019-08-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter at 30, 60 and 120 minutes after mannitol administration | 30, 60 and 120 minutes
  Change in optic nerve sheath diameter (ONSD)

SECONDARY OUTCOMES:
Correlation between change in ONSD and Mean arterial pressure | 30, 60, and 120 minutes
  Correlation with change in ONSD and Mean arterial pressure
Correlation between dose and change in ONSD | 30, 60 and 120 minutes
  Dose subgroups of <0.5gm/kg and >/= 0.5 gm/kg were compared and the correlated with changes in ONSD.

OTHER OUTCOMES:
Comparison of ONSD values among ventilated and non-ventilated patients | 30, 60 and 120 minutes
  Comparison of ONSD values among ventilated and non-ventilated patients at 30,60 and 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shiva P Paudyal, MD, Principal Investigator — Institution of medicine, Tribhuvan University, Nepal
Locations (1):
- Maharajgunj Medical Campus, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Hospital inpatient number, age, sex, weight, BMI, dose of mannitol administered, MAP, ONSD at T1, T2, T3, T4 and change in ONSD T1, T2, T3 and T4.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years
Access Criteria: Contact with the PI

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-02-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT04188353/Prot_SAP_ICF_000.pdf